CLINICAL TRIAL: NCT05300893
Title: Effectiveness of Night Splinting After Percutaneous Needle Fasciotomy in Dupuytren's Contracture - a Randomised Controlled Multicenter Trial
Brief Title: Effectiveness of Night Splinting After Percutaneous Needle Fasciotomy in Dupuytren's Contracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-01331
Record Dates: First submitted 2022-02-28; First posted 2022-03-29 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Dupuytren Contracture; Dupuytren's Disease
Keywords: Percutaneous needle fasciotomy; Splint
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with night splint after percutaneous needle fasciotomy (No Intervention)
- No treatment with night splint after percutaneous needle fasciotomy (Experimental)
  Interventions: Other: No night splint

INTERVENTIONS:
Other: No night splint — Instead of the usual treatment with a night splint for three months after percutaneous needle fasciotomy patients do not receive treatment with a night splint.
  Arms: No treatment with night splint after percutaneous needle fasciotomy

SUMMARY:
Dupuytren's contracture (DC) is associated with progressive finger flexion and extension deficit caused by fibrosis in the palm and digits. Treatment options include minimally invasive procedures such as percutaneous needle fasciotomy (PNF) and collagenase clostridium histolyticum injections as well as open fasciectomy. PNF has recently become more popular in Sweden because it is an office-based procedure which is relatively easy to perform without the usual risks and costs of open surgery.

After treatment with PNF patients usually continue with supervised rehabilitation, which includes physical therapy and night splinting. Whether night splinting is beneficial in terms of reducing recurrence of DC is currently debated.

This study aims to investigate whether night splinting after performed PNF helps to reduce recurrence rate or not. Patients who meet the inclusion criteria will be randomized into two groups: The first group will be treated as usual with physical therapy and night splinting after PNF. The second group will be treated with physical therapy without night splinting after PNF. Follow up includes physical examination regarding active range of motion, sensation and grip strength at procedure day and 2 weeks, 3, 12 and 36 months later as well as questionnaires regarding hand function, pain and quality of life at procedure day and 3, 12 and 36 months later. Patients who are randomized into the second group (no night splinting) will also be examined 3 weeks after PNF for observation in case of an early impairment regarding extension deficit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older,
* Palpable Dupuytren strand with passive extension deficit according to stadium 1 and 2 of the classification of Tubiana in one or two fingers excluding the thumb, defined as at least 30 degrees in the MCP joint and/or at least 20 degrees in the PIP joint and a maximum of 75 degrees in the MCP or PIP joint

Exclusion Criteria:

* Multiple, invasive or wide strands in the palm,
* Skin irritation,
* Strand localization in the digit only,
* Digital nerve injury,
* Any former treatment for Dupuytren's contracture in the same digit,
* Thumb contracture,
* Stadium 3 and 4 according to the classification of Tubiana

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of finger joint contracture | at 1 year follow up
  Finger joint movement in order to extend the finger measured in degrees with a goniometer before and after treatment.

SECONDARY OUTCOMES:
Change of active finger flexion | before and after treatment, at 2 weeks, 3, 12 and 36 months follow-up
  Finger joint movement in order to flex the finger measured in degrees with a goniometer before and after treatment.
Change of grip strength | before and after treatment, at 2 weeks, 3, 12 and 36 months follow-up
  The ability to grip with the hand measured with the Jamar hand dynamometer in kg before and after treatment.
Pain assessed by a numeric rating scale (NRS) | before treatment, at 3, 12 and 36 months follow-up
  Report of pain in the treated finger using a numeric rating scale from 0 to 10, where 0 is equivalent to no pain at all and 10 is equivalent to the highest thinkable pain level.
Quality of life assessed by EQ-5D | before treatment, at 3, 12 and 36 months follow-up
  Quality of life is measured by the EQ-5D questionnaire. This questionnaire is developed by the EuroQuol Group and measures 5 health dimensions: mobility, self care, usual activities, pain and discomfort, as well as anxiety and depression. The answers are transferred into an EQ-5D index from 0 to 1, where 0 is equivalent with the worst health state and 1 is equivalent with the best health state.
Dupuytren-disease-associated disability assessed by URAM | before treatment, at 3, 12 and 36 months follow-up
  The URAM (Unité Rhumatologique des Affections de la Main) scale is a 9-item questionnaire for functional assessment in Dupuytren's disease with a range from 0-45 points, where 0 is equivalent with the best functional outcome and 45 is equivalent with the worst functional outcome.
Semmes-Weinstein monofilament test | before treatment, at 3, 12 and 36 months follow-up
  Semmes-Weinstein monofilament test is a semi-quantitative test for sensory loss. Filaments in different sizes are used to put a different amount of pressure onto the skin. Depending on which filament size the patient is able to detect sensory loss can be investigated.
Study specific questionnaire concerning the patient's medical history | before treatment, at 3, 12 and 36 months follow-up
  In this questionnaire the patient answers questions about present conditions such as diabetes and smoking, therapy with pain medication for the hand, how long the patient has been diagnosed with Dupuytren'd disease, if both hands are affected and if there is a positive family history.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Wilbrand, MD, PhD, Principal Investigator — Uppsala University
Locations (3):
- Sweden (3):
  - Falu Lasarett, Falun, Dalarna County
  - Akademiska Sjukhuset, Uppsala, Uppsala County
  - Universitetssjukhuset Örebro, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-02-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT05300893/SAP_000.pdf